CLINICAL TRIAL: NCT00977119
Title: Investigation of Genetic Determinants of Capecitabine Toxicity
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: Translational Breast Cancer Research Consortium (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 09-056-B; TBCRC 015 (Other: Translational Breast Cancer Reseach Consortium)
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer
Keywords: breast cancer; capecitabine
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (including DNA)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Capecitabine: Women with breast cancer receiving capecitabine as treatment for their breast cancer.
  Interventions: Other: Side-effect questionnaires; Other: research blood samples

INTERVENTIONS:
Other: Side-effect questionnaires — Paper or telephone questionnaire to report specific side-effects associated with their breast cancer treatment weekly
Other: research blood samples — Blood samples for research on DNA before starting treatment and after 4 cycles of treatment

SUMMARY:
The purpose of this study is to identify possible genetic polymorphisms that contribute to specific toxicities associated with capecitabine (hand-foot syndrome, diarrhea, and neutropenia).

Additionally, this study will look at gene polymorphisms in patients experiencing the toxicities of interest, the frequency of polymorphisms and differences in drug metabolism.

ELIGIBILITY:
Inclusion Criteria:

* women with breast cancer in whom single agent capecitabine therapy is being considered
* aged 18 years and older

Exclusion Criteria:

* patients who have previously received capecitabine are excluded
* patients cannot be receiving capecitabine in combination with another cancer chemotherapy; concurrent use of trastuzumab is not permitted; concurrent use of zoledronic acid is allowed
* serum albumin less than 3.0 g/dL within the last 30 days
* creatinine clearance (CrCL) or glomerular filtration rate (GFR) less than 60 mL/min [/body surface area (BSA)] (within the last 30 days)
* inability to understand and give informed consent to participate
* patients with a history of inflammatory bowel disease requiring therapy or patients with chronic diarrhea syndromes or paralytic ileus
* patients with prior or concurrent pelvic irradiation
* patients who use an ostomy for fecal excretion
* there is no limit on the number of prior chemotherapies; the decision to use capecitabine is determined solely by the treating physician

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving treatment with capecitabine for breast cancer at a participating academic medical center.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2009-11-23 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Genetic variants of toxicity | 2 years

SECONDARY OUTCOMES:
Time to toxicity based on genetics | 2 years
Multiple genetic variants as predictors | 2 years
Genome-wide association (potential) | 2 years
Correlative sample collection | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter H O'Donnell, MD, Study Chair — University of Chicago
Locations (13):
- United States (13):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Georgetown University, Washington D.C., District of Columbia
  - University of Chicago, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Johns Hopkins, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University, Houston, Texas
  - M.D. Anderson Cancer Center, Houston, Texas